CLINICAL TRIAL: NCT01158703
Title: Aspirin and Plavix Following Coronary Artery Bypass Grafting (ASAP-CABG)
Brief Title: Aspirin and Plavix Following Coronary Artery Bypass Grafting
Acronym: ASAP-CABG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment and reduction in CT surgery support
Sponsor: Ahmad Slim (U.S. Federal Agency)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Slim, director, cardiovascular research, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2009.120
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Graft Patency
Keywords: aspirin; clopidogrel; coronary artery bypass graft; Plavix
MeSH Terms: interventions — Clopidogrel; Sugars; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clopidogrel (Active Comparator): aspirin and clopidogrel
  Interventions: Drug: clopidogrel; Drug: Aspirin
- sugar pill (Placebo Comparator): aspirin and placebo
  Interventions: Drug: sugar pill; Drug: Aspirin

INTERVENTIONS:
Drug: clopidogrel — clopidogrel 75mg daily by mouth daily for 12 months
  Other Names: Plavix
  Arms: clopidogrel
Drug: sugar pill — sugar pill by mouth daily for 12 months
  Other Names: placebo
  Arms: sugar pill
Drug: Aspirin — aspirin 81 mg daily by mouth for 12 months ( Standard of care in both arms)
  Other Names: ASA, acetylsalicylic acid, Ecotrin, Fasprin

SUMMARY:
The design of the study will be randomized, double blind trial, which will examine the effects of addition of clopidogrel to current guideline recommended background therapy on lowering the incidence of graft stenosis after coronary artery bypass grafting compared to placebo.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how well the combination of clopidogrel and aspirin lower the risk of clot forming in the bypass graft after open heart surgery. This combination has not yet been approved by the Food & Drug Administration (FDA) for treating clots in the bypass graft. However, the FDA has not objected to its use to study its safety and effectiveness. This study will enroll approximately 150 total subjects all of which will be at Brooke Army Medical Center/Wilford Hall Medical Center. The study will be for 52 weeks from the day of surgery.

After bypass surgery and inclusion criteria is met, subjects will be placed on aspirin 81 mg once daily and placebo once daily or aspirin 81 mg once daily and clopidogrel 75mg once daily to keep the bypass grafts open after surgery. There are no studies to date comparing the two study groups A CT scan of the heart will be done 2 weeks after surgery to see if the grafts are still open. At the end of the study, at 52-weeks mark, the subjects will undergo another heart scan to evaluate the bypass grafts and see if they are still open.

Subjects will be seen on a 3 months basis until the end of the study, unless deemed necessary to return earlier for follow up. Subjects will undergo blood draw for complete blood count as part of the follow up visits to assess for safety while on the current study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass grafting, with or without cardiopulmonary bypass
* Age ≥ 18

Exclusion Criteria:

* Left ventricle ejection fraction <30%
* Emergency surgery
* Valve surgery
* Redo CABG
* Postoperative cardiogenic shock for more than 48 hours
* Postoperative bleeding or cardiac tamponade
* More than 24 hours postoperative intubation course
* Requirement of postoperative anticoagulation
* Serum creatinine >1.4
* Contraindication to use of postoperative coronary CT scan
* Allergy or contraindication to aspirin or clopidogrel
* Inability to provide informed consent
* Pregnant or breast feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Slim, MD, Principal Investigator — Brooke Army Medical Center; Rachel Beck, MD, Study Chair — Brooke Army Medical Center; William Conner, MD, Study Chair — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clopidogrel: aspirin and clopidogrel
  clopidogrel: clopidogrel 75mg daily and aspirin 81mg by mouth daily for 12 months
- Sugar Pill: aspirin and placebo
  sugar pill: sugar pill and aspirin 81mg by mouth daily for 12 months
Period: Overall Study
Arm/Group | Clopidogrel | Sugar Pill
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two active treatment groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Sugar Pill | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.7) | 64.8 (10.2) | 66.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution among groups
  Participants
    Female | 1 | 1 | 2
    Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 117.8 (10.7) | 115.4 (12.34) | 116.8 (11.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 69.5 (9.1) | 65.1 (7.3) | 67.8 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of More Than 50% Stenosis in Graft With Combination Therapy With Aspirin and Clopidogrel vs. Aspirin Alone
Description: Incidence of more than 50% stenosis in graft with combination therapy with aspirin and clopidogrel vs. aspirin and placebo
Time Frame: 52 weeks
Population: Incidence of more than 50% stenosis in graft with combination therapy with aspirin and clopidogrel vs. aspirin and placebo
Measure: Number; unit: occluded grafts
Units Other Than Participants: grafts
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
Number analyzed (grafts) | 36 | 27
occluded grafts | 10 | 9

2. Secondary Outcome: Incidence of Bleeding Between the Two Treatment Arms
Time Frame: 52 weeks
Measure: Number; unit: BLEEDING EVENTS
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
BLEEDING EVENTS | 0 | 0

3. Secondary Outcome: Number of Major Adverse Cardiovascular Events With Combination Therapy
Description: Number of major adverse cardiovascular events(angina, any thrombotic events, and myocardial infarction) with combination therapy with aspirin and clopidogrel vs. aspirin alone
Time Frame: 52 weeks
Population: above is the total number of all events reported
Measure: Number; unit: MACE Events over 52Wks
Units Other Than Participants: All events
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
Number analyzed (All events) | 10 | 6
MACE Events over 52Wks | 10 | 6

4. Secondary Outcome: Number of Angina Events
Description: Number of angina events with combination therapy with aspirin and clopidogrel vs. aspirin alone
Time Frame: 52 weeks
Population: above is the total number of participants
Measure: Number; unit: Angina Events over 52Wks
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
Angina Events over 52Wks | 7 | 5

5. Secondary Outcome: Number of Myocardial Infarction Events
Description: Number of myocardial infarction events with combination therapy with aspirin and clopidogrel vs. aspirin alone
Time Frame: 52 weeks
Population: above is the total number of participants
Measure: Number; unit: MI Events over 52Wks
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
MI Events over 52Wks | 2 | 1

6. Secondary Outcome: Number of Thrombotic Events
Description: Number of thrombotic events with combination therapy with aspirin and clopidogrel vs. aspirin alone
Time Frame: 52 weeks
Population: above is the total number of participants
Measure: Number; unit: thrombotic Events over 52Wks
Arm/Group | Clopidogrel | Sugar Pill
Number analyzed (Participants) | 12 | 8
thrombotic Events over 52Wks | 1 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: 52 weeks events of bleeding ( TIMI Major and Minor)
Arm/Group | Clopidogrel | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 10/12 | 6/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=12) | Sugar Pill (N=8)
Number of Angina Events (Cardiac disorders) | 7 (7) | 5 (5) — Number of angina events with combination therapy with aspirin and clopidogrel vs. aspirin alone
Number of Myocardial Infarction Events (Cardiac disorders) | 2 (2) | 1 (1) — Number of myocardial infarction events with combination therapy with aspirin and clopidogrel vs. aspirin alone
Number of Thrombotic Events (Vascular disorders) | 1 (1) | 0 (0) — Number of thrombotic events with combination therapy with aspirin and clopidogrel vs. aspirin alone

LIMITATIONS AND CAVEATS:
The study did not recruit enough patients due to strict exclusion criteria and low volume of consenting patients resulting in a sample size that was insufficient for power analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No